CLINICAL TRIAL: NCT03514901
Title: An Evaluation of the Efficacy Beyond Progression of Vemurafenib Combined With Cobimetinib Associated With Local Treatment Compared to Second-line Treatment in Patients With BRAFV600 Mutation-positive Metastatic Melanoma in Focal Progression With First-line Combined Vemurafenib and Cobimetinib.
Brief Title: To Evaluate the Efficacy Beyond Progression of Vemurafenib+Cobimetinib Associated With Local Treatment Compared to Second-line Treatment in Patients With BRAFV600+ Metastatic Melanoma in Focal Progression With First-line+Vemurafenib+Cobimetinib.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Intergruppo Melanoma Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeyPro2
Record Dates: First submitted 2018-03-28; First posted 2018-05-03 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Melanoma Metastatic; BRAF V600 Mutation
MeSH Terms: interventions — pembrolizumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: A randomized, open-label study
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental combination beyond Focal Progression (Experimental): Local treatment (i.e. surgery, radiotherapy) + Vemurafenib 240mg tablets (4 tabs/twice daily for 28 consecutive days) + Cobimetinib 20mg tablets (3 tabs/day for 21 consecutive days) beyond focal progression.
  Interventions: Other: Experimental combination beyond Focal Progression
- Pembrolizumab or Nivolumab (Active Comparator): Pembrolizumab daily dose 2 mg/kg milligram(s)/kilogram or Nivolumab daily dose 3 mg/kg milligram(s)/kilogram.
  Interventions: Drug: Pembrolizumab or Nivolumab

INTERVENTIONS:
Other: Experimental combination beyond Focal Progression — Vemurafenib is taken on a 28-day cycle. Each dose consists of four 240 mg (960 mg) tablets twice daily for 28 consecutive days. The first dose should be taken in the morning and the second dose in the evening approximately 12 hours later. Each dose can be taken with or without a meal. Vemurafenib tablets should be swallowed whole with a glass of water and should not be chewed or crushed.
  Cobimetinib is taken on a 28-day cycle. Each dose consists of three 20 mg tablets (60 mg) and should be taken orally, once daily for 21 consecutive days, followed by a 7-day break. Each subsequent treatment cycle should start after the 7-day treatment break has elapsed. The dose should be taken in the morning.
  Local treatment (i.e. surgery, radiotherapy).
  Arms: Experimental combination beyond Focal Progression
Drug: Pembrolizumab or Nivolumab — Pembrolizumab 2 mg/kg is administered as an intravenous infusion over 30 minutes every 3 weeks OR Nivolumab 3 mg/kg is administered intravenously over 60 minutes every 2 weeks.
  Other Names: Keytruda or Opdivo
  Arms: Pembrolizumab or Nivolumab

SUMMARY:
The purpose of this study is to evaluate the efficacy beyond progression of vemurafenib combined with cobimetinib associated with local treatment compared to second-line treatment in patients with BRAFV600 mutation-positive metastatic melanoma in focal progression with first-line combined vemurafenib and cobimetinib.

DETAILED DESCRIPTION:
Melanoma is a heterogeneous skin tumor, characterized by mutations of different oncogenes. Almost half of patients with advanced melanoma have a gene mutation of BRAF serine-threonine kinase. Over the past 5 years, two BRAF inhibitors targeting these mutations, vemurafenib and dabrafenib, have shown high rates of rapid response in phase II and III studies. However, the duration of responses is limited in most patients due to the development of acquired resistance. Mechanisms of resistance to BRAF inhibitor therapy are diverse and include the reactivation of the mitogen-activated protein kinase (MAPK) pathway in over two-thirds of tumors, along with promotion of parallel signaling networks.

Recently, the combination of drugs was superior in terms of responses, Progression Free Survival (PFS) and Overall Survival (OS) compared to monotherapy.

The data from recent studies confirm the clinical benefit of the combination of Vemurafenib with cobimetinib and support the use of the combination as a standard first-line approach to improve survival in patients.

The aim of this randomized, open-label, phase II study is to evaluate the efficacy, in terms of overall survival, of vemurafenib combined with cobimetinib associated with local treatment compared with second-line therapy, in patients with BRAFV600 mutation-positive metastatic melanoma in focal progression with first-line combined vemurafenib and cobimetinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed melanoma, either unresectable Stage IIIc or Stage IV metastatic melanoma, as defined by the American Joint Committee on Cancer 7th edition
* Patients previously untreated for metastatic melanoma
* Documentation of BRAFV600 mutation-positive status in melanoma tumor tissue (archival or newly obtained tumor samples) by a validated mutational test
* Adequate performance status to receive vemurafenib and cobimetinib therapy as determined by treating physician
* Male or female patient aged ≥18 years
* Able to participate and willing to give written informed consent prior to any treatment-related procedures and to comply with treatment guidance
* Adequate end-organ function, defined by the following laboratory results obtained within 14 days prior to the first dose of program drug treatment:

  1. Bilirubin ≤ 1.5 x the upper limit of normal (ULN).
  2. AST, ALT, and alkaline phosphatase ≤ 3 x ULN, with the following exceptions:

     * Patients with documented liver metastases: AST and/or ALT ≤ 5 x ULN.
     * Patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 x ULN.
  3. Serum creatinine ≤1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min based on measured CrCl from a 24-hour urine collection or Cockroft-Gault glomerular filtration rate estimation.
* Female patients of childbearing potential and male patients with partners of childbearing potential must agree to always use two effective forms of contraception during program therapy and for at least 6 months after completion of program therapy
* Negative serum pregnancy test prior to commencement of dosing in women of childbearing potential
* Patient should be able to swallow tablets
* Absence of any psychological, familial, sociological, or geographical condition that potentially hampers compliance with the treatment regimen
* Patient does not currently participate in other clinical trials

Exclusion Criteria:

* Palliative radiotherapy within 7 days prior to the first dose of program treatment
* Patients with active malignancy (other than BRAF-mutated melanoma) or a previous malignancy within the past 3 years except for patients with resected melanoma, resected BCC, resected cutaneous SCC, resected melanoma in situ, resected carcinoma in situ of the cervix, and resected carcinoma in situ of the breast
* Evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment / central serous chorioretinopathy (CSCR), retinal vein occlusion (RVO), or neovascular macular degeneration
* Systemic risk factor for RVO including uncontrolled glaucoma, uncontrolled hypercholesterolemia, hypertriglyceridemia or hyperglycemia
* History of clinically significant cardiac dysfunction, including the following:

  1. Current unstable angina.
  2. Symptomatic congestive heart failure of New York Heart Association class 2 or higher.
  3. History of congenital long QT syndrome or mean (average of triplicate measurements) QTcF ≥ 450 msec at baseline; presence of clinically significant ventricular or atrial dysrhythmias ≥ Grade 2.
  4. Uncontrolled hypertension ≥ Grade 2 (patients with a history hypertension controlled with anti-hypertensives to ≤ Grade 1 are eligible).
  5. Left ventricular ejection fraction (LVEF) below institutional lower limit of normal (LLN) or below 50%, whichever is lower
* Current severe, uncontrolled systemic disease
* Major surgery or traumatic injury within 14 days prior to first dose of program treatment
* History of malabsorption or other condition that would interfere with absorption of program drugs
* Hypersensitivity to the active substance or to any of the excipients
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2023-04-29 (Estimated); Study Completion 2023-04-29 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) time for patients with focal progression | From date of randomization until the date of death from any cause, assessed up to 24 months
  Overall survival of patients with focal progression is defined as the time, in months, from randomization to the date of death from any cause. If a patient is not known to have died, survival time will be censored at the date of last contact ("last known date alive"). Overall survival of patients with focal progression will be compared between treatment groups using a log-rank test procedure with a two-sided α =0.2 level. The OS function for each treatment group will be estimated using the Kaplan-Meier product-limit method. Median and corresponding two-sided 80% confidence intervals will be computed by treatment group. A Cox proportional hazard model for OS with treatment arm as single factor will be used to estimate the hazard ratio of vemurafenib and cobimetinib plus local treatment to Standard of Care (SOC) second-line treatment and its corresponding 80% confidence interval.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) time for patients with focal progression | From date of randomization until the date of death from any cause, assessed up to 24 months
  PFS of patients with focal progression is defined as the time, in months, from randomization to the date of the first documented tumor progression or death due to any cause, whichever comes first. Clinical deterioration will not be considered progression. For subjects who neither progress nor die, time will be censored at the date of their last tumor assessment. For subjects who start a new anti-tumor treatment, time will be censored at the start of the new treatment. For a randomized subject who does not have any post-randomization tumor assessments and who has not died, time will be censored at the randomization date. PFS will be compared between treatment groups using a log-rank test procedure with a two-sided α =0.2 level. The PFS function for each treatment group will be estimated using the Kaplan-Meier product-limit method. Median and two-sided 80% confidence intervals (CI) for median PFS will be computed by treatment group. A Cox proportional hazard model for PFS with treatment
Overall Survival (OS) time for patients with non-focal progression | From date of the last dose of vemurafenib and cobimetinib until the date of death from any cause, assessed up to 24 months
  Overall survival of patients with non-focal progression is defined as the time, in months, from date of non-focal progression to first-line to the date of death from any cause. If a patient is not known to have died, survival time will be censored at the date of last contact ("last known date alive"). The OS function will be estimated using the Kaplan-Meier product-limit method. Median and corresponding two-sided 80% confidence intervals will be computed. Overall survival results of patients with non-focal progression will be descriptively compared with OS results of patients with focal progression (i.e. primary efficacy endpoint).
Comparison between Overall Survival (OS) time for patients with non-focal progression and Overall Survival (OS) results of patients with focal progression | From date of randomization or date of the last dose of vemurafenib and cobimetinib until the date of death from any cause, assessed up to 24 months
  Overall survival results of patients with non-focal progression will be descriptively compared with OS results of patients with focal progression (i.e. primary efficacy endpoint). No statistical test will be foreseen for this comparison. The overall survival results are defined as the time, in months, from the date of progression to the date of death.
Nature of adverse events (AE) and serious adverse events (SAE) reported throughout the study | From baseline up to 24 months after the last treatment
  Nature of adverse events (AE) and serious adverse events (SAE) verified during the study. Safety analyses will be reported by actual treatment group and on the Non-focal Progression Set. AE and SAE will be assessed according to the Common Terminology Criteria for AEs (CTCAE version 4).
Frequency of adverse events (AE) and serious adverse events (SAE) reported throughout the study | From baseline up to 24 months after the last treatment
  Frequency of adverse events (AE) and serious adverse events (SAE) verified during the study. Safety analyses will be reported by actual treatment group and on the Non-focal Progression Set. AE and SAE will be assessed according to the Common Terminology Criteria for AEs (CTCAE version 4).
Severity of adverse events (AE) and serious adverse events (SAE) reported throughout the study | From baseline up to 24 months after the last treatment
  Severity of adverse events (AE) and serious adverse events (SAE) verified during the study. Safety analyses will be reported by actual treatment group and on the Non-focal Progression Set. AE and SAE will be assessed according to the Common Terminology Criteria for AEs (CTCAE version 4).
Timing of adverse events (AE) and serious adverse events (SAE) reported throughout the study | From baseline up to 24 months after the last treatment
  Timing of adverse events (AE) and serious adverse events (SAE) verified during the study. Safety analyses will be reported by actual treatment group and on the Non-focal Progression Set. AE and SAE will be assessed according to the Common Terminology Criteria for AEs (CTCAE version 4).
Changes in blood pressure | From baseline up to 24 months
  Changes in blood pressure during and following vemurafenib + cobimetinib administration. Blood pressure will be measured in mmHg (millimetres of mercury).
Changes in heart rate | From baseline up to 24 months
  Changes in heart rate during and following vemurafenib + cobimetinib administration. Heart rate will be measured in bpm (beats per minute).
Changes in temperature | From baseline up to 24 months
  Changes in temperature during and following vemurafenib + cobimetinib administration. Temperature will be measured in °C (degrees centigrade).
Changes in respiratory rate | From baseline up to 24 months
  Changes in respiratory rate during and following vemurafenib + cobimetinib administration. Respiratory rate will be measured in breaths per minute.
Changes in clinical laboratory results | From baseline up to 24 months
  Changes in clinical laboratory results during and following vemurafenib + cobimetinib administration. Laboratory results will be assessed according to the Common Terminology Criteria for AEs (CTCAE version 4).

CONTACTS AND LOCATIONS:
Overall Officials: Paola Queirolo, Dr., Principal Investigator — Ospedale Policlinico San Martino di Genova
Locations (14):
- Italy (14):
  - Istituto dei Tumori "Giovanni Paolo II", Bari, BA
  - ASST Papa Giovanni XXIII, Bergamo, BG
  - Policlinico Sant'Orsola Malpighi, Bologna, BO
  - IRCCS IRST Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, FC
  - Ospedale Policlinico San Martino, Genova, GE
  - P.O. di Taormina - Azienda Sanitaria Provinciale di Messina, Taormina, ME
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - Istituto Oncologico Veneto - IRCCS, Padua, PD
  - Ospedale S. Chiara - A.O.U. Pisana, Pisa, PI
  - A.O.U.S. Policlinico "Le Scotte", Siena, SI
  - P.O. San Lazzaro - A.O.U. Città della Salute e della Scienza di Torino - Molinette, Torino, TO
  - Istituto Europeo di Oncologia - Divisione Melanoma, Sarcoma e Tumori Rari, Milan
  - Istituti Fisioterapici Ospitalieri - IFO - Istituto "Regina Elena", Roma
  - IDI Istituto Dermopatico Immacolata, Roma

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT03514901/Prot_SAP_000.pdf